CLINICAL TRIAL: NCT03161652
Title: Clinical Trial to Evaluate the Safety and Efficacy of Levosulpiride to Improve Retinal Alterations in Patients With Diabetic Retinopathy and Diabetic Macular Edema.
Brief Title: Effect of Levosulpiride on Retinal Alterations in Patients With Diabetic Retinopathy and Diabetic Macular Edema
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carmen Clapp (Other)
Collaborators: Instituto Mexicano de Oftalmologia (IMO) (Unknown); Universidad Autónoma de Querétaro (Other); General Hospital Nuremberg & Paracelsus Medical University Nuremberg (Unknown); Instituto de la Retina del Bajio SC (INDEREB) (Unknown); Instituto de Neurobiología, Universidad Nacional Autonoma de Mexico (UNAM) (Unknown)
Responsible Party: Sponsor-Investigator, Carmen Clapp, Principal Investigator, Universidad Nacional Autonoma de Mexico
Organization: Universidad Nacional Autonoma de Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDRDME_247164
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: diabetic retinopathy; blindness; eye; macular edema; prolactin; dopamine antagonists; peptide hormones
MeSH Terms: conditions — Diabetic Retinopathy; Blindness; Macular Edema | interventions — Sugars; dimethylethylsilylimidazole

STUDY DESIGN:
Intervention Model Description: The study investigates a medication causing hyperprolactinemia (levosulpiride) to treat diabetic retinopathy (DR) and diabetic macular edema (DME). Subjects are from four different populations, those with DME, non-proliferative DR, those undergoing vitrectomy due to proliferative DR, and those with DME plus standard intravitreal antiangiogenic therapy with ranibizumab. Immediately after baseline, each of the four groups are randomly split into two subgroups: one receiving placebo (sugar pill) and the other levosulpiride. Ophthalmologic and health outcomes between groups 1 and 2 (DME: placebo and levosulpiride), 3 and 4 (DR: placebo and levosulpiride), and 7 and 8 (DME plus ranibizumab: placebo and levosulpiride) evaluate the efficacy and safety of the study medication. Comparison of serum and vitreous prolactin levels between the groups undergoing vitrectomy (DR: placebo and levosulpiride) serve as a proof of principle that prolactin enters the eye to counteract disease progression.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, care providers, and evaluators are blind to treatment allocation. This reduces the risk of bias in the measurement of outcomes, in the decision to modify or discontinue treatment, or to withdraw from trial or from analysis. The monitoring coordinator allocates the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- DME lactose pill (Placebo Comparator): Patients with DME will be randomized to take a lactose pill (placebo).
  Interventions: Drug: DME lactose pill
- DME levosulpiride (Experimental): Patients with DME will be randomized to take levosulpiride.
  Interventions: Drug: DME levosulpiride
- DR lactose pill (Placebo Comparator): Patients with non-proliferative DR will be randomized to take a lactose pill (placebo)
  Interventions: Drug: DR lactose pill
- DR levosulpiride (Experimental): Patients with non-proliferative DR will be randomized to take levosulpiride
  Interventions: Drug: DR levosulpiride
- DR, vitrectomy lactose pill (Placebo Comparator): Patients with proliferative DR (undergoing medically prescribed vitrectomy 7 days after starting the study) will be randomized to take a lactose pill (placebo).
  Interventions: Drug: DR vitrectomy lactose pill
- DR, vitrectomy levosulpiride (Experimental): Patients with proliferative DR (undergoing medically prescribed vitrectomy 7 days after starting the study) will be randomized to take levosulpiride.
  Interventions: Drug: DR vitrectomy levosulpiride
- DME plus ranibizumab lactose pill (Placebo Comparator): Patients with DME that will receive intravitreal antiangiogenic therapy with ranibizumab will be randomized to take a lactose pill (placebo)
  Interventions: Drug: DME plus ranibizumab lactose pill
- DME plus ranibizumab levosulpiride (Experimental): Patients with DME that will receive intravitreal antiangiogenic therapy with ranibizumab will be randomized to take levosulpiride
  Interventions: Drug: DME plus ranibizumab levosulpiride

INTERVENTIONS:
Drug: DME lactose pill — Patients with DME will take placebo orally 3 times a day (TID) for 8 weeks.The placebo is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: placebo, sugar
  Arms: DME lactose pill
Drug: DME levosulpiride — Patients with DME will take levosulpiride (75 mg/day) orally TID for 8 weeks. Levosulpiride is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: dopamine D2 receptor blocker
  Arms: DME levosulpiride
Drug: DR lactose pill — Patients with non-proliferative DR will take a lactose pill (placebo) orally TID for 8 weeks. The placebo is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: placebo, sugar
  Arms: DR lactose pill
Drug: DR levosulpiride — Patients with non-proliferative DR will take levosulpiride (75 mg/day) orally TIDfor 8 weeks. Levosulpiride is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: dopamine D2 receptor blocker
  Arms: DR levosulpiride
Drug: DR vitrectomy lactose pill — Patients with proliferative DR (undergoing medically prescribed vitrectomy 7 days after starting the study medication) will have to take a lactose pill (placebo) orally TID for one week. The last placebo pill will be taken on the morning of the day vitrectomy is performed. The placebo is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: placebo, sugar
  Arms: DR, vitrectomy lactose pill
Drug: DR vitrectomy levosulpiride — Patients with proliferative DR (undergoing medically prescribed vitrectomy 7 days after starting the study medication) will take levosulpiride (75 mg/day) orally TID for one week. The last pill will be taken on the morning of the day vitrectomy is performed. Levosulpiride is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: dopamine D2 receptor blocker
  Arms: DR, vitrectomy levosulpiride
Drug: DME plus ranibizumab lactose pill — Patients with DME with conventional intravitreal antiangiogenic therapy with ranibizumab (0.5 mg every 4 weeks for 12 weeks) will take a lactose pill (placebo) orally TID for 24 weeks. The placebo is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: placebo, sugar
  Arms: DME plus ranibizumab lactose pill
Drug: DME plus ranibizumab levosulpiride — Patients with DME with receive intravitreal antiangiogenic therapy with ranibizumab (0.5 mg every 4 weeks for 12 weeks) will take a levosulpiride (75 mg/day) orally TID for 24 weeks. The study medication is taken on top of standard therapy for diabetes and blood pressure control.
  Other Names: dopamine D2 receptor blocker
  Arms: DME plus ranibizumab levosulpiride

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of levosulpiride to improve retinal alterations due to diabetic macular edema and diabetic retinopathy

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) and diabetic macular edema (DME) are the primary cause of irreversible blindness and visual impairment in working-age adults. Nearly 80% of patients with diabetes will experience some degree of DR and DME 15-20 years after diagnosis. Altered blood parameters (glucose, lipids, and pressure) influence disease development and progression; however, the combined values of these parameters account for only 10% of the risk of DR. Laser therapy is effective for preserving sight but is poor for reversing visual loss. Anti-angiogenic therapies are effective and less destructive but require frequent intravitreal delivery, which raises the risk of infection and ocular complications. Therefore, the prevention and treatment of DR and DME should include other modifiable factors. Data from preclinical studies support a protective role for the serum levels of the hormone prolactin. The trial investigates a new specific therapy for DR and DME based on elevating the circulating levels of prolactin with the prokynetic, dopamine D2 receptor blocker, levosulpiride. It is a prospective, randomized clinical study in patients with DR and DME in which ophthalmologic and health parameters evaluated before and after starting the study medication will determine the efficacy and safety of treatment.

Patient registries: Patients are enrolled at the time of a routine health care service. The caregiver and patient together, in a standardized uniform manner for every patient, will collect the data. Data collection procedures are clearly described and include protocols, policies, and the formatted listing of all the data elements, their full definitions and validation rules. All personnel involved in data collection are qualified registry trained. The same physicians, laboratory technicians, and graduate students will evaluate and collect the data from all patients. An individual fully knowledgeable of all protocols, policies, procedures, and definitions in the registry will be designated as Accountable for Data Quality. This individual (coordinator) should ensure that all collected data are complete, accurate, and valid. Data logically inconsistent will be confronted to information in external database. Data collected on formatted paper forms are entered into a computer and electronic registries carefully reviewed by a third party to identify missing data, invalid or erroneous entries, and inconsistent data. Any data review activity and remediation efforts will be documented. Amelioration of data problems may include querying the personnel uploading the data, the coordinator, the interviewer, or the patient. The proposed sample size and study duration are the minimum required and are based on biological models of DR and on clinical experience evaluating primary data associated with the study. These parameters may have to be modified to accommodate the sample size required to obtain clinically important differences and their statistical evaluation, access to eligible patients, lack of adherence to therapy at specific calendar dates (holidays), etc. Statistical methods include those evaluating continuous and categorical variables, incidence and prevalence, the association between a risk factor and outcome, and the relative contribution of confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 40 years but no older than 69 years
* Male and female subjects with mild and moderate diabetic macular edema (DME), non-proliferative diabetic retinopathy (DR), and with proliferative DR undergoing medically prescribed vitrectomy.
* Signing informed consent
* Without ocular complications: severe myopia (> 6 diopters), ocular media opacity, retinal detachment, etc.
* Without previous ocular treatments: ocular surgeries, retinal laser photocoagulation, intravitreal administration of antiangiogenic agents (delivered < 6 months before enrollment).
* Prolactin serum levels ≤ 20 ng/ml
* With normal or mild loss of kidney function (glomerular filtration rate >60 ml/min) for groups with DME and DR without vitrectomy.
* With mild to severe loss of kidney function (glomerular filtration rate >30 ml/min) for groups with DR undergoing vitrectomy.
* Without contraindications for the use of levosulpiride (Parkinson disease, epilepsy, breast cancer, alcoholism, hypokalemia).
* Without hyperprolactinemia inducing conditions: Pathologies (hypothyrodism, hepatic dysfunction, prolactinomas); Medication (antipsychotics, antidepressants, prokinetics, other)

Exclusion Criteria:

* Not meeting inclusion criteria.
* Adverse and intolerable drug effects.
* Not complying with study medication
* Inability to continue in-hospital appointments.
* Missing outcome data
* Hesitation to continue with study medication
* Relocation to another state or country
* Voluntary withdrawal of consent

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 5 minutes
  Number of letters recognized in the Early Treatment Diabetic Retinopathy Study (ETDRS) chart test after correcting for any refractive error (myopia, hyperopia, or astigmatism)
Retinal thickness | Pupils are dilated (eye drops) for 10 to 15 minutes and optical coherence tomography (OCT) images recorded during 5 minutes.
  Retinal thickness is evaluated by non-invasive optical coherence tomography (OCT) imaging via qualitative and quantitative analyses. For qualitative analyses, OCT images approaching the histological level of retinal morphology are interpreted based on normal and diseased features (hyper-reflective or hypo-reflective lesions, shadowing, and anatomical changes). Quantitative analysis evaluates retinal reflective signals and their correlation with retinal morphology by computer image-processing algorithms (retinal thickness map, volume, area, 1, 3, and 6 mm ETDRS circle diameters).
Retinal hard exudates and hemorrhages | Pupils are dilated (eye drops) for 10 to 15 minutes and fundus images recorded during 5 minutes
  Number, size, and location of retinal hard exudates and hemorrhages evaluated by indirect ophthalmoscopy
Retinal microaneurisms, leakage area, cotton-wool spots, venous beading, microvascular and vascular abnormalities | Pupils are dilated (eye drops) for 10 to 15 minutes and fundus images recorded before and at different times (0.5 to 5 minutes) after fluorescein injection.
  Location, intensity, and source of above alterations evaluated by fundus fluorescein angiography imaging qualitative and quantitative analysis of hyper-fluorescent or hypo-fluorescent regions.
Prolactin serum levels | 1-2 minutes (duration of blood withdrawal)
  ng/ml levels of prolactin quantified in serum samples using the IMMULITE 2000 XPi immunoassay system
Prolactin vitreous levels | 2 minutes (duration of vitreous withdrawal during medically prescribed vitrectomy)
  ng/ml levels of prolactin quantified in vitreous samples using the IMMULITE 2000 XPi immunoassay system
Vasoinhibin vitreous levels | 2 minutes (duration of vitreous withdrawal during medically prescribed vitrectomy)
  Optical density values of vasoinhibins obtained by the immunoprecipitation-Western blot analysis of vitreous samples

SECONDARY OUTCOMES:
Pyruvic glutamic transaminase (TGP) and thyroid stimulating hormone (TSH) serum levels | 1-2 minutes (duration of blood withdrawal)
  U/L (TGP) and uU/mL (TSH) quantified in serum samples by the Bioclin Kinetic Transaminase ALT (TGP) Kit and the automatic quimioluminescent evaluator (TSH)
Blood glycated hemoglobin and creatinine serum levels | 1-2 minutes (duration of blood withdrawal)
  Glycated hemoglobin (evaluated by boronate affinity chromatography) and creatinine (evaluated by the Jaffe reaction) levels are expressed as % and mg/dL, respectively.
Blood pressure | 5 minutes
  Systolic and diastolic values in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Clapp, Ph.D., Study Director — Universidad Nacional Autonoma de Mexico (UNAM); Ludivina Robles Osorio, M.D., Ph.D., Principal Investigator — Universidad Autónoma de Querétaro; Renata Garcia Franco, M.D., Principal Investigator — Instituto de la Retina del Bajio SC (INDEREB); Jakob Triebel, M.D., Principal Investigator — Institute for Clinical Chemistry, Laboratory Medicine and Transfusion Medicine, Nuremberg General Hospital; Marlon R Garcia Roa, M.D., Principal Investigator — Instituto Mexicano de Oftalmología (IMO)
Locations (2):
- Mexico (2):
  - Instituto Mexicano de Oftalmologia (IMO), Querétaro City, Querétaro
  - Instituto de la Retina del Bajio SC (INDEREB), Querétaro City, Querétaro

IPD SHARING:
Plan to Share IPD: Undecided
It is yet undecided whether case reports will be published in medical journals throughout the course of the study. No identifier linking participants in the study to research records will be made public or reported.

REFERENCES:
- [Background] Aranda J, Rivera JC, Jeziorski MC, Riesgo-Escovar J, Nava G, Lopez-Barrera F, Quiroz-Mercado H, Berger P, Martinez de la Escalera G, Clapp C. Prolactins are natural inhibitors of angiogenesis in the retina. Invest Ophthalmol Vis Sci. 2005 Aug;46(8):2947-53. doi: 10.1167/iovs.05-0173. PMID 16043870
- [Background] Garcia C, Aranda J, Arnold E, Thebault S, Macotela Y, Lopez-Casillas F, Mendoza V, Quiroz-Mercado H, Hernandez-Montiel HL, Lin SH, de la Escalera GM, Clapp C. Vasoinhibins prevent retinal vasopermeability associated with diabetic retinopathy in rats via protein phosphatase 2A-dependent eNOS inactivation. J Clin Invest. 2008 Jun;118(6):2291-300. doi: 10.1172/JCI34508. PMID 18497878
- [Background] Clapp C, Thebault S, Arnold E, Garcia C, Rivera JC, de la Escalera GM. Vasoinhibins: novel inhibitors of ocular angiogenesis. Am J Physiol Endocrinol Metab. 2008 Oct;295(4):E772-8. doi: 10.1152/ajpendo.90358.2008. Epub 2008 Jun 10. PMID 18544641
- [Background] Arnold E, Rivera JC, Thebault S, Moreno-Paramo D, Quiroz-Mercado H, Quintanar-Stephano A, Binart N, Martinez de la Escalera G, Clapp C. High levels of serum prolactin protect against diabetic retinopathy by increasing ocular vasoinhibins. Diabetes. 2010 Dec;59(12):3192-7. doi: 10.2337/db10-0873. Epub 2010 Sep 7. PMID 20823101
- [Background] Triebel J, Macotela Y, de la Escalera GM, Clapp C. Prolactin and vasoinhibins: Endogenous players in diabetic retinopathy. IUBMB Life. 2011 Oct;63(10):806-10. doi: 10.1002/iub.518. Epub 2011 Sep 13. PMID 21913303
- [Background] Ramirez M, Wu Z, Moreno-Carranza B, Jeziorski MC, Arnold E, Diaz-Lezama N, Martinez de la Escalera G, Colosi P, Clapp C. Vasoinhibin gene transfer by adenoassociated virus type 2 protects against VEGF- and diabetes-induced retinal vasopermeability. Invest Ophthalmol Vis Sci. 2011 Nov 21;52(12):8944-50. doi: 10.1167/iovs.11-8190. PMID 22003113
- [Background] Arnold E, Thebault S, Baeza-Cruz G, Arredondo Zamarripa D, Adan N, Quintanar-Stephano A, Condes-Lara M, Rojas-Piloni G, Binart N, Martinez de la Escalera G, Clapp C. The hormone prolactin is a novel, endogenous trophic factor able to regulate reactive glia and to limit retinal degeneration. J Neurosci. 2014 Jan 29;34(5):1868-78. doi: 10.1523/JNEUROSCI.2452-13.2014. PMID 24478366
- [Background] Arredondo Zamarripa D, Diaz-Lezama N, Melendez Garcia R, Chavez Balderas J, Adan N, Ledesma-Colunga MG, Arnold E, Clapp C, Thebault S. Vasoinhibins regulate the inner and outer blood-retinal barrier and limit retinal oxidative stress. Front Cell Neurosci. 2014 Oct 20;8:333. doi: 10.3389/fncel.2014.00333. eCollection 2014. PMID 25368550
- [Background] Diaz-Lezama N, Wu Z, Adan-Castro E, Arnold E, Vazquez-Membrillo M, Arredondo-Zamarripa D, Ledesma-Colunga MG, Moreno-Carranza B, Martinez de la Escalera G, Colosi P, Clapp C. Diabetes enhances the efficacy of AAV2 vectors in the retina: therapeutic effect of AAV2 encoding vasoinhibin and soluble VEGF receptor 1. Lab Invest. 2016 Mar;96(3):283-95. doi: 10.1038/labinvest.2015.135. Epub 2015 Nov 16. PMID 26568297
- [Background] Melendez Garcia R, Arredondo Zamarripa D, Arnold E, Ruiz-Herrera X, Noguez Imm R, Baeza Cruz G, Adan N, Binart N, Riesgo-Escovar J, Goffin V, Ordaz B, Pena-Ortega F, Martinez-Torres A, Clapp C, Thebault S. Prolactin protects retinal pigment epithelium by inhibiting sirtuin 2-dependent cell death. EBioMedicine. 2016 May;7:35-49. doi: 10.1016/j.ebiom.2016.03.048. Epub 2016 Apr 20. PMID 27322457
- [Background] Robles-Osorio ML, Garcia-Franco R, Nunez-Amaro CD, Mira-Lorenzo X, Ramirez-Neria P, Hernandez W, Lopez-Star E, Bertsch T, Martinez de la Escalera G, Triebel J, Clapp C. Basis and Design of a Randomized Clinical Trial to Evaluate the Effect of Levosulpiride on Retinal Alterations in Patients With Diabetic Retinopathy and Diabetic Macular Edema. Front Endocrinol (Lausanne). 2018 May 29;9:242. doi: 10.3389/fendo.2018.00242. eCollection 2018. PMID 29896154
- See also: Carmen Clapp's research web page — http://personal.inb.unam.mx/clapp/
- See also: Instituto de Neurobiologia, Universidad Nacional Autonoma de Mexico web page — http://www.inb.unam.mx/
- See also: Instituto Mexicano de Oftalmologia web page — https://imoiap.com.mx/